CLINICAL TRIAL: NCT02677207
Title: The Effects of JNJ-39393406 on Psychometric Performance and Residual Depressive Symptoms in 80 Patients With Unipolar or Bipolar Depression: a Phase II Exploratory add-on Double Blind Placebo Controlled 2 Week Trial
Brief Title: The Effects of JNJ-39393406 on Psychometric Performance and Residual Depressive
Acronym: JNJ-DEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tangent Data (Other)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JNJ-DEP
Record Dates: First submitted 2016-01-21; First posted 2016-02-09 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2018-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — JNJ-39393406

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-39393406 (Experimental): 2 capsules, once daily for the first week and 4 capsules once a day for the rest of the trial.
  Interventions: Drug: JNJ-39393406
- Placebo (Placebo Comparator): 2 capsules, once daily for the first week and 4 capsules once a day for the rest of the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-39393406 — JNJ-39393406 100 mg capsules or placebo daily for the first week and 200 mg daily for the rest of the trial
  Arms: JNJ-39393406
Drug: Placebo — JNJ-39393406 100 mg capsules or placebo daily for the first week and 200 mg daily for the rest of the trial
  Arms: Placebo

SUMMARY:
To evaluate the effects of the nicotinic allosteric modulator JNJ-39393406 on psychometric performance and residual depressive symptoms in patients who have been diagnosed with unipolar and bipolar depression but currently DO NOT meet criteria for an episode of Major Depression or Manic Episode.

DETAILED DESCRIPTION:
To evaluate the effects of the nicotinic allosteric modulator JNJ-39393406 on psychometric performance and residual depressive symptoms in patients who have been diagnosed with unipolar and bipolar depression but currently DO NOT meet criteria for an episode of Major Depression or Manic Episode.

Hypothesis: Allosteric modulation of the a7nAChR with JNJ-39393406 improves psychometric performance and residual depressive symptoms in patients with unipolar major depression disorder (MDD) or bipolar depression (BPD).

Outcome measurements:

* BACS
* MADRS
* BNSS
* CGI-S- BP,
* Questionnaire on smoking urges (QSU) and time to the first cigarette after waking up in the morning,
* Readiness for discharge scale.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM V criteria for history of MDD or BPD by MINI.
2. Between 18-50 years of age, male or female subjects of any race, smokers and non-smokers.
3. Able to provide informed consent. All participant patients must have signed an informed consent document indicating they understand the purpose of the study and the procedures required for the study and are willing to participate by complying with the study procedures and restrictions.
4. Have a MADRS ≥ 10 and ≤ 34 and an YMRS < 7.
5. In the opinion of the investigator, basic education and severity of symptoms (psychotic, negative, manic, agitation, depression) do not prevent the patient from attending to the cognitive tasks.
6. In the opinion of the investigator the patient can be safely treated with no more than 2 psychotropic medications as background therapy (SOS for agitation and sleeping medication are allowed in addition to the 2 psychotropics).
7. The background psychotropic(s) that will be continued through-out the 2 week trial must have been started at least 2 weeks prior to the baseline day at doses allowed by the local regulations and no changes in dose have been made during this pre-baseline 2 week period.
8. Inpatients or out-patients at the discretion of the investigator (If outpatients the Readiness for Discharge Scale has to be administered at baseline and at each visit.)

Exclusion Criteria:

1. Women of child bearing potential who do not practice contraception.
2. Psychosis, florid manic or major depressive episode during the 4 weeks preceding baseline day or current psychosis.
3. Patients on more than 2 psychotropic (hypnotics for sleep and occasional SOS for agitation do not count).
4. Smokes more than 40 cigarettes per day.
5. Unstable medical disease (malignancy, poorly controlled diabetes, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning. Particular attention should be given to exclude patients with ischemic heart disease).
6. Has a clinically significant abnormal 12-lead electrocardiogram (ECG) at Screening Visit 1 as determined by the Investigator.
7. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
8. Patients with a current DSM-V substance or alcohol dependence.
9. Concurrent delirium, mental retardation, drug-induced psychosis, or history of stroke, brain degenerative disorders and brain trauma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of the nicotinic allosteric modulator JNJ-39393406 on cognition | two weeks - each study visit
  Brief Assessment of Cognition (BACS)

SECONDARY OUTCOMES:
To evaluate the effects of JNJ-39393406 on depressive symptoms | two weeks - each study visit
  Montgomery-Asberg Depression Scale (MADRS)
To evaluate the effects of JNJ-39393406 on residual depressive symptoms | two weeks - each study visit
  Brief Negative Symptoms Scale (BNSS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, M.D., Principal Investigator — Principal Investigator
Locations (4):
- Clinical Psychiatric Hospital, Codru, Moldova
- Romania (3):
  - S.C. Stefi-Dent Srl, Botoșani
  - Hospital of Psychiatry and Neurology, Brasov
  - Spit. Clinic de Urgenta Militar "Dr. Stefan Odobleja", Craiova

IPD SHARING:
Plan to Share IPD: Yes